CLINICAL TRIAL: NCT01929161
Title: Affective and Genomic Mediators of Sustained Behavior Change: A Randomized, Dual-blind, Placebo-controlled Experimental Design That Will Examine Wellness Behavior as a Function of Oxytocin vs. Placebo.
Brief Title: Study of Wellness Behaviors as a Function of Oxytocin vs Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Barbara L. Fredrickson, PhD, Kenan Distinguished Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 12-2371 IRB; R01NR012899-03S2 (NIH)
Record Dates: First submitted 2013-08-01; First posted 2013-08-27 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Sustained Positive Emotions; Sustained Positive Behavior Change
Keywords: positive emotions; meditation; oxytocin
MeSH Terms: interventions — Oxytocin; Mindfulness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oxytocin (Experimental): Oxytocin intranasal spray, 6 intranasal sufflations which deliver a total of 24 international units of oxytocin
  Interventions: Drug: Oxytocin; Behavioral: Lovingkindness Meditation; Behavioral: Mindfulness Meditation
- Placebo (for oxytocin) (Placebo Comparator): Intranasal spray with all equivalent ingredients except oxytocin
  Interventions: Drug: Placebo (for oxytocin); Behavioral: Lovingkindness Meditation; Behavioral: Mindfulness Meditation
- Lovingkindness Meditation (Experimental): Lovingkindness guided meditation experienced in the laboratory and 6 additional LKM meditations taken home on the iPod.
  Interventions: Drug: Oxytocin; Drug: Placebo (for oxytocin); Behavioral: Lovingkindness Meditation
- Mindfulness Meditation (Placebo Comparator): Mindfulness guided meditation experienced in the laboratory and 6 additional Mindfulness meditations taken home on the iPod.
  Interventions: Drug: Oxytocin; Drug: Placebo (for oxytocin); Behavioral: Mindfulness Meditation

INTERVENTIONS:
Drug: Oxytocin — 24 International Units
  Other Names: Syntocinon
  Arms: Lovingkindness Meditation; Mindfulness Meditation; Oxytocin
Drug: Placebo (for oxytocin) — intranasal spray manufactured to mimic oxytocin nasal spray
  Arms: Lovingkindness Meditation; Mindfulness Meditation; Placebo (for oxytocin)
Behavioral: Lovingkindness Meditation
  Arms: Lovingkindness Meditation; Oxytocin; Placebo (for oxytocin)
Behavioral: Mindfulness Meditation
  Arms: Mindfulness Meditation; Oxytocin; Placebo (for oxytocin)

SUMMARY:
The specific aim of this study is to test whether oxytocin (OT) boosts the positive emotion yield of a new wellness behavior (Lovingkindness meditation or Mindfulness meditation) and thereby increases nonconscious motives that shape daily behavioral decisions to repeat it, which in turn foster positive emotions that further augment nonconscious motives in an upward spiral dynamic.

The proposed research targets three hypotheses: (1) Oxytocin manipulation magnifies (i.e., moderates) the positive emotion yield of Lovingkindness meditation; (2) The positive emotion yield of meditation, which varies by experimental condition, increases the nonconscious incentive salience of Wellness Behavior-related cues; and (3) Behavioral decisions predict positive emotions, sparking the relationships among OT manipulation, positive emotion yield, and nonconscious incentive salience of Wellness Behavior-related cues.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 35 and 64 years old.
* Fluent in written and spoken English
* Willingness or interest in learning to meditate
* Computer literate with access to internet (weekly)

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Individuals on antihypertensive medication
* Individuals who have or have had a regular meditation practice
* Individuals who can read Chinese logographs

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in positive emotions (as measured by the Modified Daily Emotions Scale) | Baseline and Weeks 1, 2, and 3
  Modified Daily Emotions Scale (mDES) - This measure of explicit positive affect has been successfully used by the PI in multiple studies to detect changes in positive emotion. Previous work by the PI found that Cronbach's alpha coefficient for the mDES positive emotion composite variable was 0.93 in sample of mid-life community adults similar to those anticipated for this study.
Change in nonconscious incentive salience (as measured by the Affect Misattribution Procedure). | Baseline and Weeks 1, 2, and 3
  Affect Misattribution Procedure (AMP) - This measure of nonconscious incentive salience has acceptable internal consistency for an indirect measure of affect (.69 - .90) and has been found to predict judgments and behavioral outcomes above and beyond self-report measures.
Changes in meditation time | Weeks 1, 2, and 3
  Self-reported meditation time recorded daily and weekly. In addition, meditation track play times will be recorded from the iPod.

SECONDARY OUTCOMES:
Cardiac Vagal Tone | Baseline
  This measure of parasympathetic control over the heart has been positively associated with both emotional and social functioning. Previous work by the PI's team has found that baseline vagal tone predicts increased positive response to lovingkindness meditation (LKM), and that LKM in turn increases vagal tone. Previous research by other labs has also found that OT administration increases vagal reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Fredrickson, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC PEP Lab, Chapel Hill, North Carolina, United States